CLINICAL TRIAL: NCT01441570
Title: The Impact of Nebivolol Versus Metoprolol on Quality of Life Measures and Cost-effectiveness in Stable Renal Transplant Recipients
Brief Title: The Impact of Nebivolol Versus Metoprolol on Quality of Life
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to slow enrollment
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Forest Laboratories (Industry); Lahey Clinic (Other)
Responsible Party: Principal Investigator, Steven Gabardi, Abdominal Organ Transplant Specialist, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011P001638
Record Dates: First submitted 2011-09-26; First posted 2011-09-27 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-03

CONDITIONS: Transplant; Failure, Kidney; Hypertension
Keywords: kidney; transplant; hypertension; nebivolol; metoprolol; bystolic; toprol
MeSH Terms: conditions — Hypertension | interventions — Nebivolol; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nebivolol (Active Comparator)
  Interventions: Drug: Nebivolol
- Metoprolol Succinate (Active Comparator)
  Interventions: Drug: Metoprolol succinate

INTERVENTIONS:
Drug: Nebivolol — Subject will take nebivolol daily for 12 weeks.
  Other Names: Bystolic
  Arms: Nebivolol
Drug: Metoprolol succinate — Subject will take metoprolol succinate daily for 12 weeks.
  Other Names: Toprol XL
  Arms: Metoprolol Succinate

SUMMARY:
In an open label analysis, nebivolol has been shown to have a positive impact on quality of life in the general hypertensive population. That is, patients treated with nebivolol reported less side effects compared to those treated with metoprolol. Also, more nebivolol treated patients reached normalization of blood pressure. Although there is no data, it is believed that the impact would be similar in renal transplant recipients.

The primary goal of this study is to determine if nebivolol will improve the quality of life measurements of kidney transplant recipients as compared to those treated with metoprolol succinate. This will be measured by comparing the scores of four quality of life questionnaires taken before and after 12 weeks of treatment with study drug. Other aims of this study are to determine if the use of nebivolol is cost-effective in the renal transplant recipient; determine if there is a change in urine protein excretion and renal function with the use of nebivolol; and determine the number of patients that maintain or achieve a target blood pressure of ≤ 120/80 mmHg.

ELIGIBILITY:
Inclusion Criteria:

* Adult renal transplant recipients, men and women between 18 and 75 years of age, inclusive.
* Patients must be > 3 months post-transplant.
* Patients must have stable renal function (stable renal function will be defined as those patients without infection or hospitalization [for any reason] over the past 30 days, and patients with < 20% change in their serum creatinine over the past 30 days.
* Patients receiving corticosteroids must be receiving a daily dose of < 7.5 mg of prednisone (or therapeutic equivalents based on glucocorticoid equivalency scale).
* All eligible patients must be receiving antihypertensive medication management which must include metoprolol tartrate or metoprolol succinate.
* Patients may be on more than one medication to control their hypertension. Use of any other FDA-approved antihypertensive agent is permitted.
* All eligible patients will either be at goal blood pressure (<120/80 mmHg) or have Pre-hypertension (<140/90 mmHg) or Stage I hypertension (<160/100 mmHg) at the time of study inclusion.
* Patients who are able to comprehend and satisfactorily comply with protocol requirements.
* Patients who signed the written informed consent given prior to entering any study procedure.

Exclusion Criteria:

* Patients with Stage II/uncontrolled hypertension (>159/99 mmHg).
* Patients with an easily identifiable etiology for fatigue (i.e. anemia, iron-deficiency, poor sleep patterns, etc.).
* Patients who have a medical condition that, in the Investigator's opinion, would expose them to an increased risk of a significant adverse event or interfere with assessments of safety and efficacy during the course of the trial (i.e. arrhythmia).
* Patients with any current malignancy, or any clinically significant hematological, endocrine, cardiovascular, hepatic, gastrointestinal or neurological disease (including any form of epilepsy). If there is a history of such disease but the condition has been stable for at least the past year and is judged by the investigator not to interfere with the patient's participation in the study, the patient may be included.
* Patients who are judged by the investigator to be unable or unlikely to follow the study protocol and complete all scheduled visits.
* Patients with any contraindications to beta blocker therapy as listed in the package labeling for both metoprolol succinate and nebivolol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Gabardi, PharmD, FCCP, BCPS, Principal Investigator — Transplant Surgery
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nebivolol | Metoprolol Succinate
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebivolol | Metoprolol Succinate | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life
Description: Primary outcome measure will be the change from the Screening/Enrollment Visit to the End of the Study/Early Termination visit in scores of four quality of life questionnaires. The four quality of life questionnaires that were used included the following:
  1. Short Form (SF)-36v2 Health Survey (Score Range = 0-100; the lower the score the more disability)
  2. Sexual Dysfunction Tool for Men = International Index of Erectile Function (IIEF) Questionnaire (Score Range = 5-25; a score of 22-25 = No erectile dysfunction; 17-21 = Mild erectile dysfunction; 12-16 = Mild to moderate erectile dysfunction; 8-11 = Moderate erectile dysfunction; 5-7 = Severe erectile dysfunction)
  3. Sexual Dysfunction Tool for Women = Changes in Sexual Functioning Questionnaire (CSFQ-14-F; Score Range = 14-70; a score at or below 42 is indicative of sexual dysfunction)
  4. Multidimensional Assessment of Fatigue (MAF) Scale (Score Range = 1-50; the higher the score the more fatigue)
Time Frame: 12 weeks; Baseline scores were measured at the Initial Screening/Enrollment Visit (Visit 1 - beginning of week 1); Follow-Up scores were measured at the End of the Study (Visit 2 - End of week 12)
Population: Adult (>18 years of age) renal transplant recipients, both men and women, requiring pharmacotherapy for high blood pressure were evaluated for inclusion in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Metoprolol: Metoprolol succinate: Subject will take metoprolol succinate daily for 12 weeks.
Arm/Group | Nebivolol | Metoprolol
Number analyzed (Participants) | 6 | 5
units on a scale
  Baseline SF-36 (physical) Score | 41.1 (5.3) | 45.9 (13.3)
  Follow-Up SF-36 (physical) Score | 46.6 (13.6) | 43.6 (15.1)
  Change from Baseline SF-36 (physical) | 5.5 (10.1) | -2.3 (8.4)
  Baseline SF-36 (mental) Score | 40.6 (12) | 40.3 (11.1)
  Follow-Up SF-36 (mental) Score | 48 (11.7) | 42.7 (13.3)
  Change from Baseline SF-36 (mental) | 7.4 (8) | 2.4 (7.1)
  Baseline MAF Score | 27.7 (8.3) | 31.7 (8.6)
  Follow-Up MAF Score | 22.1 (12.2) | 17.8 (12.2)
  Change from Baseline MAF | -5.6 (6.3) | -13.9 (9.1)
  Baseline IIEF Score | 10.3 (15.3) | 15 (9.8)
  Follow-Up IIEF Score | 16.3 (14.6) | 14.3 (12.3)
  Change from Baseline IIEF | 6.7 (9.9) | -1.3 (0.6)
  Baseline CSFQ | 48.7 (0.6) | 49 (0)
  Follow-Up CSFQ | 53.0 (5.7) | 49 (0)
  Change from Baseline CSFQ | 4.5 (6.4) | 0 (0)

2. Secondary Outcome: Blood Pressure
Description: Evaluate the baseline and follow-up systolic and diastolic blood pressures for all subjects in both groups.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Nebivolol | Metoprolol
Number analyzed (Participants) | 6 | 5
mmHg
  Baseline Systolic Blood Pressure | 142.3 (14.6) | 138.8 (14.3)
  Follow-Up Systolic Blood Pressure | 142.8 (10.7) | 136.0 (13.9)
  Change from Baseline Systolic Blood Pressure | 3.6 (8.9) | -2.8 (9.9)
  Baseline Diastolic Blood Pressure | 73.2 (8.5) | 77.0 (9.9)
  Follow-Up Diastolic Blood Pressure | 76.0 (5.7) | 73.0 (13.7)
  Change from Baseline Diastolic Blood Pressure | 1.6 (4.8) | -4.0 (11.2)

ADVERSE EVENTS:
Arm/Group | Nebivolol | Metoprolol
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No